CLINICAL TRIAL: NCT02859753
Title: Prospective Randomized Controlled Study Comparing Response and Recurrence Rates Following Percutaneous Microwave Coagulation Therapy (MCT) Versus Percutaneous Radiofrequency Ablation (RFA) in Patients With Chronic Liver Disease and Hepatocellular Carcinoma
Brief Title: Comparison of Response and Recurrence Rates Following Percutaneous Microwave Coagulation Therapy Versus Percutaneous Radiofrequency Ablation
Acronym: Thermoablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GUIU MicroS 2012
Record Dates: First submitted 2016-08-01; First posted 2016-08-09 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Thermoablation; Chronic Liver Disease; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Catheter Ablation

ARMS (2):
- RFA (Experimental)
  Interventions: Other: Percutaneous Radiofrequency Ablation
- MCT (Active Comparator)
  Interventions: Other: Percutaneous Microwave Ablation

INTERVENTIONS:
Other: Percutaneous Radiofrequency Ablation
  Arms: RFA
Other: Percutaneous Microwave Ablation
  Arms: MCT

SUMMARY:
To date, the majority of studies that have evaluated the efficacy of microwave ablation (MWA) in the treatment of hepatocellular carcinoma (HCC) lesions in cirrhotic patients and compared its efficacy with that of percutaneous radiofrequency ablation (RFA) for local recurrence and survival have been retrospective. There have been no prospective randomized studies comparing percutaneous microwave ablation (PMWA) with RFA for ablated tumour volume, the response after one session, local recurrence rates in the first year, complication rates and survival at 3 and 5 years for HCC lesions > 2 cm in patients with Child-Pugh A and B cirrhosis. The hypothesis the investigators wish to explore is that though the 2 methods are equivalent for lesions ≤ 2 cm, MWA could show better efficacy with a similar risk for lesions > 2 cm and for lesions close to vessels ≥ 3 mm in diameter, as shown in retrospective studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient who have been informed about the research and given their oral consent
* Patients with national health insurance cover
* Patients ≥ 18 years
* ≤ 3 CHC lesions ≤ 4 cm, with a maximum of 3 lesions with a diagnosis of HCC based on histology, or according to European Society for the Study of the Liver (EASL) criteria
* Chronic liver disease or cirrhosis with a Child-Pugh score between 5 and 8 points
* Contra-indication for surgical resection at the time of the therapeutic decision made during a multidisciplinary meeting

Exclusion Criteria:

* Informed consent not obtained (refusal of patient or patient lacking discernment)
* Kidney failure with creatinine clearance < 30 ml/min thus preventing the injection of contrast for the initial or follow-up radiological imaging
* Presence of a malignant tumour other than the HCC at the time of the diagnosis, unless a basocellular carcinoma
* Cirrhosis with a Child-Pugh score > 8
* Contra-indication for percutaneous treatment according to Barcelona Clinic Liver Cancer (BCLC) criteria
* Patients without national health insurance cover

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-01-15 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Time to disease progression according to American Society of Interventional Radiology criteria | Through study completion up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Derived] Vietti Violi N, Duran R, Guiu B, Cercueil JP, Aube C, Digklia A, Pache I, Deltenre P, Knebel JF, Denys A. Efficacy of microwave ablation versus radiofrequency ablation for the treatment of hepatocellular carcinoma in patients with chronic liver disease: a randomised controlled phase 2 trial. Lancet Gastroenterol Hepatol. 2018 May;3(5):317-325. doi: 10.1016/S2468-1253(18)30029-3. Epub 2018 Mar 2. PMID 29503247